CLINICAL TRIAL: NCT02445833
Title: Design, Development And Validation Of A On-Line Intervention For Promoting Healthy Habits And Weight Loss In Hypertensive And Risk For Diabetes Mellitus People With Overweight And Type I Obesity
Brief Title: On-Line Intervention For Promoting Healthy Habits And Weight Loss In Hypertensive Patients
Acronym: VIVIR-MEJOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: University of Valencia (Other); Cardenal Herrera University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vivir mejor
Record Dates: First submitted 2015-04-22; First posted 2015-05-15 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Obesity
Keywords: Obesity; Internet intervention; Cardiovascular disease; Hypertension; Lifestyle intervention; Weight loss treatment
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle on-line intervention (Experimental): The self-applied on-line intervention will received acces to the web and the "Vivir mejor" modules.
  Interventions: Behavioral: Lifestyle on-line intervention

INTERVENTIONS:
Behavioral: Lifestyle on-line intervention — The self-applied on-line intervention will comprise a behavioural intervention composed by 9 modules seeking to develop gradually achieving the goals of changing eating habits and physical activity in participants (Themes: 1.motivation for change; 2. nutrition and physical activity education; 3. barriers to change, healthy eating principles and how to be active; 4. Influence of thoughts; 5. Emotional eating and self-control; 6. Problem solving; 7. Body image and assertiveness; 8. Relapse prevention)..The program will be established as follows: The first day the participant log in the website where can access the processing modules. A web page was developed specially for this study.
  Other Names: VIVIR MEJOR

SUMMARY:
Efficacy of an Internet-based self-guided intervention for promoting healthy habits and weight loss in hypertensive people with overweight and obesity: A Randomized Controlled Trial

DETAILED DESCRIPTION:
The prevalence of overweight and obesity is on the rise worldwide with severe physical and psychosocial consequences. Hypertension is one of the comorbidities associated with obesity. Changes in lifestyles through eating behavior and physical activity level are the critical components in the prevention and treatment for hypertension and obesity. Data from several studies indicate that the usual procedures to promote these healthy habits in health services are inadequate. ICTs has been demonstrated as an effective tool for implementation of psychological interventions focused on this type of population. This study aims to describe a totally self-applied online program (¨Vivir Mejor¨) to promote healthy lifestyles (eating behavior and physical activity) for obese participants with hypertension. Participants (BMI=25-35) will be recruited from users of a hypertension unit of a public hospital and will be randomized into two groups: experimental group "Vivir Mejor" and control group (treatment as usual). "Vivir Mejor" program is composed by 9 modules aimed for promoting healthy eating habits and increase physical activity. Modules will be sent via Internet periodically. After 6 months, a follow-up testing phase and a tracking module will be set. The outcomes variables will include anthropometric data, changes in eating behavior and physical performance and cardiovascular variables.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese grade I (BMI> 25 and <35)
* Age between 18-65 years
* Being in clinical medical treatment for prevention of metabolic syndrome or Cardiac complications
* Having internet access.

Exclusion Criteria:

* No Internet access; Taking more than 3 antihypertensive drugs
* Have Diabetes diagnosis; Meet the DSM-IV-TR of Eating Disorder
* Submit a serious psychological disorder diagnosed (psychosis, bipolar disorder, major depressive disorder, substance abuse)
* Have a disability which prevents or hinders the exercise and physical activity
* Be receiving any treatment for weight loss in another center.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes in blood pressure levels at 6 and 12 months | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  (arterial brachial systolic and diastolic pressure, determined by Omron®; in millimeters of mercury)

SECONDARY OUTCOMES:
Quality of life variables with the Quality of life-QLI | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  Quality of life-QLI (Mezzich, Cohen and Ruiperez 1999; Spanish version of Mezzich et al, 2000): It includes 10 items, with multiple-choice Likert response format, consisting of a scale of 1 to 10. Evaluates 10 areas: physical, psychological, self-care and independent functioning welfare, occupational functioning , interpersonal functioning, social-emotional support, community and support services, personal fulfillment, spiritual fulfillment, overall perception of quality of life.
Food Intake style with Dutch Eating Behaviour Questionnaire | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  DEBQ- Dutch Eating Behavior Questionnaire (Van Strien et al, 1986). Translated into Spanish by Baños, 2011): Evaluates styles posing contribute intake or attenuate the development of overweight. It is composed of 33 items, with Likert scale of 5 points.
Pyshical activity with the International Physical Activity Questionnaire - IPAQ - short | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  - International Physical Activity Questionnaire - IPAQ - short (Booth, 2000.): Self-report of 7 items that collects information about PA and sedentary behavior of people in four areas: activity at work, when traveling, at home and during leisure time (leisure). The IPAQ addresses the number of days and minutes for performing physical activities such as leisure-time occupations, locomotion and housework activities. The score is derived from the number of days, hours and minutes employed therein (Carral & Perez, 2011).
Self-efficacy with the Self-Efficacy Questionnaire General | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  GSES-12 Self-Efficacy Questionnaire General (Baessler & Schwarcer, 1996): Self-report scale consisting of 10 items with Likert scales of 4 points. It was designed to assess the overall efficacy and evaluates the stable sense of personal competence to effectively manage a variety of stressful situations
Regulation of behavior in physical exercise and eating habits with BREQ-2 | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  BREQ-2 - Scale regulation of behavior in physical exercise and eating habits (Markland & Tobin, 2004. Validated to the Spanish context by Moreno, Cervellò & Martinez Camacho, 2006): The original questionnaire was developed to measure external regulation, introjected, identified and intrinsic motivation. The BREQ-2 scale consists of 19 items, compared with 15 of the original scale, measuring stages of the continuum of self-determination. An adaptation of this scale also be conducted to assess motivation to change eating habits.
Blood preasure | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  Pressure Arterial brachial systolic and diastolic (determined by Omron®; in millimeters of mercury), Central systolic and diastolic blood pressure (measured by MOBIL-O-GRAPH®; augmentation index), speed of the pulse wave; Afectación By vascular arterial stiffness parameters: speed of the pulse wave (PWV) and analysis of the pulse wave, augmentation index and central arterial pressure (measured by oscillometric brachial (MOBIL-O-GRAPH®) and carotid distensibility ultrasound (ESAOTE®);
Estimation Indirect fitness level / activity energy expenditure using portable accelerometer (Actigraph GT1M®) | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  To assess cardiorespiratory endurance test subjects performed the 6MWT (Test of 6-minute walk): cardiorespiratory functional test consists of measuring the maximum distance you can go walking a subject for 6 minutes. In each participant the routes meters, average heart rate (MHR) during test development (monitored through digital heart rate monitor Polar 610si®) and heart rate recovery phase to post-minute effort was recorded (FCR1 );
Body Mass Index | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  (Body Mass Index = kilograms / height 2(meters).
Satisfaction with treatment | It will be avaluated before and after a 3 months intervention, and follow up in 6 and 12 months.
  6-item scale with a 10-point Likert scale. It evaluates the user's opinion about the program received in terms of satisfaction and usefulness.

REFERENCES:
- [Derived] Banos RM, Mensorio MS, Cebolla A, Rodilla E, Palomar G, Lison J, Botella C. An internet-based self-administered intervention for promoting healthy habits and weight loss in hypertensive people who are overweight or obese: a randomized controlled trial. BMC Cardiovasc Disord. 2015 Aug 4;15:83. doi: 10.1186/s12872-015-0078-1. PMID 26239241